CLINICAL TRIAL: NCT06892353
Title: AI-powered Low-cost Portable Fundus Camera to Deliver Diabetic Retinopathy Screening At Primary Health Care Setting: a Pragmatic Trial
Brief Title: AI-Powered DIY Screening System for Diabetic Retinopathy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: HSEARS20231218003
Record Dates: First submitted 2025-02-07; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-02

CONDITIONS: Diabetic Retinopathy
Keywords: diabetic retinopathy; AI; screening system
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Screening (Experimental): All the participants will undertake an AI-powered fundus camera screening, physician/optometrist consultation, survey with questionnaires and a phone interview three months after their baseline assessment.
  Interventions: Diagnostic Test: AI-powered fundus camera screening

INTERVENTIONS:
Diagnostic Test: AI-powered fundus camera screening — All the participants will undertake an AI-powered fundus camera screening, physician/optometrist consultation, survey with questionnaires and a phone interview three months after their baseline assessment.

SUMMARY:
A pragmatic trial will be conducted in two representative clinics in each of the three types of targeted settings. It will be run for 3 months in each clinic to complete data collection of up to 100 patients in SPGC and Optometry Clinics, 200 at GPGC and 200 in GOPC in total. All the subjects will conduct a DIY screening, physician consultation, survey with questionnaires and a phone interview three months after their baseline assessment. This study will assess automated screening in terms of success rate of the DIY system without active assistant help, accuracy, screening rate and detection rate, adherence to referral and experience of participants, as well as cost-effectiveness in real-world settings.

ELIGIBILITY:
Inclusion Criteria:

1. subjects who are 50 years of age or older, or subjects who are 18 years of age or older and have diabetes, and
2. have not undertaken an eye examination in the previous 12 months (elevated risk of undiagnosed disease).
3. Provide written informed consent.

Exclusion Criteria:

1. individuals with physical disabilities that prevent the use of a fundus camera, or
2. individuals with speech impairments who are unable to complete telephone follow-ups.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Success Rate without Active Assistant Help | 3 months
  Success rate of using the DIY screening booth help will be determined by the number of successful screening runs without active assistant help divided by the total number of screening runs.

SECONDARY OUTCOMES:
Assessment of Consumer Acceptability | 3 months
  Assessment of consumer acceptability will be determined by the positive response rate/screening rate (i.e. the total number of eligible patients who agree to screening (numerator) divided by the total number of eligible individuals (denominator)).
Diagnostic Accuracy | 3 months
  All retinal images will be re-graded by two independent ophthalmologists, with any disagreements adjudicated by a third ophthalmologist (gold standard). This grading result will be considered as gold standard reference for the diagnostic accuracy of the automated screening. The indicators for diagnostic accuracy include: sensitivity.
Disease Detection Rates | 3 months
  The detection rate is defined as the proportion of newly diagnosed DR cases divided by the total number of eligible individuals.
Adherence to Referral | 3 months
  Patient adherence to referral will be measured as the proportion of patients who attend an ophthalmology service among the total number of referred patients.
Technical Feasibility: Quality of Image Acquisition | 3 months
  The investigators will use a standardized checklist to assess the quality of images acquired during the study. This checklist will include criteria resolution, clarity, and completeness of the images. A sample of images will be reviewed by a panel of experts to ensure consistency and reliability in the assessment.
Cost-effectiveness of DIY Screening | 3 months
  The cost-effective analyses will involve using the incremental cost-effectiveness ratio (ICER) as the key indicator to identify whether DIY screening model is a good investment.
Assessment of Consumer Satisfaction | 3 months
  The responses to the 5-point Likert scale question will be analysed using the "document variable statistics" function in MAXQDA software. Data from the open-ended questionnaire will be analysed thematically. All themed information will be shared for review by project steering committee. The Likert scale ranges from 1 to 5. The content includes 5 options, including strongly disagree, disagree, neural, agree, strongly agree. The higher scores (e.g., 4 or 5) indicate a stronger agreement or a more positive attitude towards the statement, while lower scores (e.g., 1 or 2) indicate disagreement or a more negative attitude.
Diagnostic Accuracy | 3 months
  All retinal images will be re-graded by two independent ophthalmologists, with any disagreements adjudicated by a third ophthalmologist (gold standard). This grading result will be considered as gold standard reference for the diagnostic accuracy of the automated screening. The indicators for diagnostic accuracy include: specificity.
Diagnostic Accuracy | 3 months
  All retinal images will be re-graded by two independent ophthalmologists, with any disagreements adjudicated by a third ophthalmologist (gold standard). This grading result will be considered as gold standard reference for the diagnostic accuracy of the automated screening. The indicators for diagnostic accuracy include: accuracy.
Diagnostic Accuracy | 3 months
  All retinal images will be re-graded by two independent ophthalmologists, with any disagreements adjudicated by a third ophthalmologist (gold standard). This grading result will be considered as gold standard reference for the diagnostic accuracy of the automated screening. The indicators for diagnostic accuracy include: positive/negative predictive values.
Diagnostic Accuracy | 3 months
  All retinal images will be re-graded by two independent ophthalmologists, with any disagreements adjudicated by a third ophthalmologist (gold standard). This grading result will be considered as gold standard reference for the diagnostic accuracy of the automated screening. The indicators for diagnostic accuracy include: area under curve.
Technical Feasibility:The duration of Clinic Flow | 3 months
  The investigators will conduct time-motion studies to evaluate the impact of the new imaging process on clinic flow. This will track the time taken for image acquisition, processing, and reporting and record the total time spent.
Technical Feasibility:Reporting and Impact on Clinic Flow | 3 months
  The investigators will involve track any delays or disruptions in the clinic schedule.
Technical Feasibility: The type of technical error | 3 months
  The investigators will maintain a log of technical errors encountered during the image acquisition process. This log will include the type of error.
Technical Feasibility: Number of Recorded Technical Errors | 3 months
  The investigators will maintain a log of technical errors encountered during the image acquisition process. This log will record the frequency of each type of technical errors.
Technical Feasibility: Remedies for technical errors | 3 months
  The investigators will maintain a log of technical errors encountered during the image acquisition process. This log will document any corrective actions taken in response to technical errors. Regular review meetings will be held to analyze these errors and implement strategies to minimize their occurrence.

CONTACTS AND LOCATIONS:
Locations (1):
- SPGC and Optometry Clinics, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No